CLINICAL TRIAL: NCT02899481
Title: Role of Intrapartum Ultrasound in the Efficacy of an Instrumental Delivery
Brief Title: Role of Intrapartum Ultrasound in Instrumental Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data Safety Monitoring Committee recommended stopping the trial due to futility.
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Joana Barros, MD, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-157
Record Dates: First submitted 2016-07-06; First posted 2016-09-14 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group will be constituted by pregnant women in whom the operative delivery will be preceded by a transabdominal and transperineal ultrasound to evaluate fetal head position and fetal head station, by means of determination of the 'angle of progression'.
  Interventions: Other: Transabdominal and transperineal ultrasound
- Control group (No Intervention): The control group will be constituted by pregnant women in whom the operative delivery will be carried out based solely on clinical criteria, namely transvaginal digital examination.

INTERVENTIONS:
Other: Transabdominal and transperineal ultrasound — Transabdominal ultrasound, for determining fetal head position, is performed with the pregnant women in supine position after bladder emptying, with the transducer placed transversely on the suprapubic region of the maternal abdomen. For the sonographic determination of the fetal descent we will perform a transperineal ultrasound achieved by placing the ultrasound transducer on the perineum in a mid sagittal position between the labia below the pubic symphysis.
  Arms: Study group

SUMMARY:
Investigators will perform a multicentric randomized controlled trial comparing the effect of transabdominal and transperineal ultrasound in pregnant women in the second stage of labor, in whom it was decided an operative delivery. Our objective is to evaluate the impact of intrapartal ultrasound measurements, as an auxiliary to clinical evaluation, in the efficacy of an instrumental delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term, in labor (≥ 37 weeks of gestation dated by a first trimester ultrasound
* live singleton pregnancy
* fetus in a cephalic presentation
* in the second stage of labor, after the decision to perform an instrumental delivery

Exclusion Criteria:

* fetal malformations
* emergency situation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Maternal and neonatal morbidity | 2 years
  Severe postpartum hemorrhage, perineal trauma, prolonged hospital stay
Neonatal morbidity | 2 years
  low 5-minute Apgar score, umbilical artery metabolic acidosis, birth trauma and neonatal intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Joana Barros, MD, Principal Investigator — University of Lisbon
Locations (1):
- Centro Hospitalar Lisboa Norte - Hospital Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No